CLINICAL TRIAL: NCT03433391
Title: Confirmatory Clinical Study to Support the Effectiveness and Safety of Oxiplex for the Reduction of Pain and Symptoms Following Lumbar Surgery
Brief Title: Confirmatory Clinical Study of Oxiplex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FzioMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FZ-SP007
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Herniated Lumbar Disk

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Surgery Plus Oxiplex (Other): Oxiplex will be applied after hemostasis is achieved and prior to closure, in adult patients undergoing single level partial discectomy.
  Interventions: Device: Oxiplex
- Surgery Only (Other): Standard of care procedures for adult patients undergoing single level partial discectomy will be followed.
  Interventions: Other: Surgery Only

INTERVENTIONS:
Device: Oxiplex — Oxiplex is a clear, viscoelastic gel that is applied to operative site during lumbar spine surgery in order to coat the nerve root with a protective barrier.
  Arms: Surgery Plus Oxiplex
Other: Surgery Only — Single level partial discectomy as per standard of care procedures.
  Arms: Surgery Only

SUMMARY:
This is a prospective, multi-center, randomized, controlled, patient and evaluator-blinded clinical study to assess the safety and effectiveness for the reduction of pain and symptoms following lumbar surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Be between 22 and 70 years of age;
2. Have symptomatic posterior or posterolateral disc herniation at L4-L5 or L5-S1 with radiographic confirmation of nerve compression using MRI that requires partial surgical discectomy with or without laminotomy;
3. Have radiculopathy (e.g., decreased motor strength, sensory deficits, decreased reflexes) from specific nerve root distribution from L4 to S1 with positive straight leg raise (0-60 degrees);
4. Have at least one of the following:

   1. At least six weeks of prior conservative treatment (e.g., physical therapy and/or use of anti-inflammatory medications, narcotics, and muscle relaxants at the manufacturer's recommended therapeutic dose);
   2. The patient is experiencing intractable pain; or
   3. There is substantial progression of loss of neurological function.
5. Have VAS leg pain score in the ipsilateral leg of at least 60mm on a 100mm scale;
6. Have VAS back pain score of at least 50mm on a 100mm scale;
7. Be appropriate for treatment using a posterior surgical approach;
8. Be likely to return for all follow-up visits; and
9. Be willing and able to provide Informed Consent for study participation.

Exclusion Criteria:

Pre-Operative Exclusion Criteria:

1. Radiographic confirmation (via MRI) of severe facet disease or facet degeneration at the index lumbar level;
2. Prior spine surgery at any lumbar level;
3. Subject requires spinal surgery other than a partial discectomy (with or without laminotomy) to treat leg/back pain (osteophyte removal is allowed);
4. Previous trauma to the lumbar spine resulting in fracture or documented ligament injury;
5. Documented presence of a free nuclear fragment at lumbar levels other than the study level;
6. Axial back pain only (no radicular symptoms);
7. Recent history (within previous six months) of chemical or alcohol dependence;
8. Active systemic infection;
9. Infection at the site of surgery;
10. Cauda equina syndrome or neurogenic bowel/bladder dysfunction;
11. Any terminal, systemic or autoimmune disease;
12. Metabolic bone disease (e.g., osteoporosis/osteopenia, gout, osteomalacia, Paget's disease); as defined by use of anti-resorptive medications or a history of fragility fracture;
13. Any disease, condition or surgery which might impair healing, such as:

    * Diabetes mellitus requiring daily insulin management,
    * Active malignancy,
    * History of metastatic malignancy;
14. Treatment with any epidural steroids within four (4) weeks prior to the surgery;
15. Treatment with any oral steroids within ten (10) days prior to the surgery;
16. Treatment with aspirin or other non-steroidal anti-inflammatory drugs within seventy-two (72) hours prior to the surgery;
17. Currently experiencing an episode of major mental illness (psychosis, major affective disorder, or schizophrenia), or manifesting physical symptoms without a diagnosable medical condition to account for the symptoms, which may indicate symptoms of psychological rather than physical origin;
18. Pregnancy at time of enrollment, or planning to become pregnant, since this would contraindicate surgery2;
19. Currently a prisoner;
20. Currently involved in litigation which may influence the subject's reporting of symptoms including workers comp;
21. Participation in any other investigational drug, biologic or medical device study within the last six months prior to study surgery;
22. Requires removal of far lateral disc herniations at L4/5 or L5/S1.

Intra-operative Exclusion Criteria:

In case the surgeon identifies during surgery any circumstance that contradicts to the patient's participation in the trial, the surgeon should exclude the patient from trial participation. Exclusion reasons are:

1. Severe facet disease or facet degeneration at the index lumbar level;
2. Dural entry during surgery;
3. Discovery of intraspinal tumor during surgery;
4. Requires spinal fusion;
5. Multilevel herniation or the need to involve more than one level;
6. Exploration of contralateral side;
7. Epidural fat placement;
8. Application of products to the exposed neural element, including:

   * Amniotic tissue or fluids
   * Adhesives
   * Steroids
   * Platelet rich plasma
   * Gelfoam
   * Allograft tissue
   * Fibrin glue
   * Dural patches
9. Surgical determination that a hemostatic agent must remain at the surgery site;
10. Surgical determination of the need for any other device (that would interfere with interpretation of the study results) to remain at the surgery site (e.g., surgical drains);
11. Adverse events or complications assessed during surgery that rule out the use of Oxiplex (e.g., infection, local osteoporosis);
12. Application of a sealant or other attempt to repair annular tear;
13. Implantation of antibiotic powder into the surgical wound. (Antibiotic irrigation may be used in the treatment group prior to Oxiplex application and the control group following surgery. No irrigation is allowed after Oxiplex application.);
14. The presence of a dural tear and/or opening found during the surgical procedure.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Change in ipsilateral leg pain | Pre-op; 6 weeks; 3 months; 6 months
  Subjects will complete a Visual Analogue Scale (VAS) for their ipsilateral leg pain at each visit. The VAS is a continuous and linear, scale ranging from "No Pain" to "Worst Possible Pain".

SECONDARY OUTCOMES:
Change in back pain | Pre-op; 6 weeks; 3 months; 6 months
  Subjects will complete a Visual Analogue Scale (VAS) for their back pain at each visit.The VAS is a continuous and linear, scale ranging from "No Pain" to "Worst Possible Pain".

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Fischgrund, MD, Principal Investigator — Beaumont Health
Locations (17):
- United States (17):
  - Desert Institute for Spine Care, Phoenix, Arizona
  - Center for Neurosciences, Tucson, Arizona
  - UC Davis Spine Center, Sacramento, California
  - Kennedy-White Orthopaedic Center, Sarasota, Florida
  - Orlando Neurosurgery, Winter Park, Florida
  - Rush University Medical Center, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Indiana Spine Group, Carmel, Indiana
  - Orthopaedic Institute of Western Kentucky, Paducah, Kentucky
  - Brigham and Women's Hospital, Boston, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - St. Luke's Hospital, Kansas City, Missouri
  - Northwell Health Physician Partners, Great Neck, New York
  - OrthoCarolina Research Insitute, Charlotte, North Carolina
  - M3 Emerging Medical Research, Durham, North Carolina
  - Texas Back Institute, Plano, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rhyne AL, Blumenthal SL, Frank EH, Hsu KY, Kim KD, Youssef JA, Wang JC, Arnold P, BenDebba M, Block KM, Juarez TG, Chiacchierini RP, Ehmsen RJ, Krelle JS, diZerega GS; Oxiplex Clinical Study Group. Oxiplex reduces leg pain, back pain, and associated symptoms after lumbar discectomy. Spine (Phila Pa 1976). 2012 Apr 15;37(8):631-41. doi: 10.1097/BRS.0b013e3182309af7. PMID 21897344
- [Background] Kim KD, Wang JC, Robertson DP, Brodke DS, Olson EM, Duberg AC, BenDebba M, Block KM, diZerega GS. Reduction of radiculopathy and pain with Oxiplex/SP gel after laminectomy, laminotomy, and discectomy: a pilot clinical study. Spine (Phila Pa 1976). 2003 May 15;28(10):1080-7; discussion 1087-8. doi: 10.1097/01.BRS.0000062354.26905.B8. PMID 12768153
- See also: Sponsor Website — http://www.fziomed.com/